CLINICAL TRIAL: NCT07354919
Title: A Phase II Trial of Cancer Response Using Axelopran in Patients With Advanced Cancers on Opioids (AxeCan)
Brief Title: Axelopran in Advanced Cancers
Acronym: AxeCan
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Glycyx MOR Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AxeCan
Record Dates: First submitted 2026-01-19; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Lung Cancer; Pancreas Cancer; Prostate Cancer
Keywords: cancer; axelopran; opioids
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axelopran monotherapy (Experimental): axelopran capsules administered daily as monotherapy
  Interventions: Drug: axelopran

INTERVENTIONS:
Drug: axelopran — axelopran capsules

SUMMARY:
The primary objective of this single arm, open label, phase II trial is to determine if axelopran use impacts cancer control in patients with advanced cancers of the lung, breast, pancreas, and prostate. The primary study period for assessing the primary aim is through day 43 (6 weeks). The main questions it aims to answer are:

* Does axelopran show a signal for efficacy in slowing tumor progression?
* Is axelopran safe and tolerable for long-term use in this patient population?
* Does axelopran show a signal for efficacy in improving bowel function and quality of life?
* Does axelopran show a signal for efficacy in reducing systemic inflammation, cachexia, and prognostic serum biomarkers of inflammation?

Patients will take axelopran as monotherapy after relapse or progression on or after standard systemic therapy. Clinician and patient must be willing to attempt a delay in next line of systemic cancer therapy (if available) until day 43 to assess change in cancer status on repeat imaging. Clinician can move to the next line of therapy whenever deemed clinically necessary.

Participants will:

* take oral axelopran capsules daily for up to 1 year, or longer if deriving benefit
* attend 10 in-person study visits, each lasting approximately 1-2 hours
* complete study procedures including but not limited to imaging exams, blood draws, electronic health surveys, and physical assessments

ELIGIBILITY:
Inclusion Criteria:

1. Adults (aged 18 or more at enrollment).
2. Histologically or cytologically proven cancer of the prostate (carcinoma), breast (carcinoma), pancreas (carcinoma), and lung (non-small cell lung carcinoma (NSCLC)) that has relapsed or progressed on or after a standard systemic treatment that has included cytotoxic chemotherapy.
3. Advanced stage (locally advanced or metastatic) with no definitive plans for curative-intent therapy.
4. A minimum life expectancy of at least 2 months at the time of the screening visit.
5. Current use of an opioid medication with an average of 5mg OME/day over the past 3 days.
6. At least one measurable lesion meeting RECIST v1.1 criteria.
7. At least 2 weeks since last cancer-directed therapy:

   1. NSCLC and pancreatic cancer must have received at least one line of systemic cytotoxic chemotherapy (+/- immune checkpoint inhibitor) in the locally advanced/metastatic setting.
   2. Breast cancer must be considered hormone-refractory and have received at least one line of systemic cytotoxic chemotherapy in the locally advanced/metastatic setting.
   3. Prostate cancer must be considered metastatic castrate-resistant prostate cancer (mCRPC) and have progressed on at least one androgen receptor pathway inhibitor (ARPI) and docetaxel. Docetaxel could be given in the metastatic castrate-sensitive setting, and/or later in the mCRPC setting. Baseline testosterone level must be <50 ng/dL and surgical or ongoing medical castration must be maintained throughout the duration of the study.
8. Patients must a) have relapsed or progressed on or after all standard therapy, b) be intolerant to standard therapy, c) not have standard therapy available that confers a significant clinical benefit, d) decline other standard therapy or agree with treating oncologist that a period of active surveillance off therapy is reasonable.
9. Clinician and patient are willing to attempt a delay in next line of systemic cancer therapy (if available) until day 43 to assess change in cancer status on repeat imaging. Clinician can move to next line of therapy at any time if a patient's clinical course changes and urgent new treatment is required. Patients will be allowed to remain on axelopran if that occurs.

   a) Planned palliative radiation therapy should be completed prior to study enrollment. Palliative radiation done during the primary study period would be considered next line of cancer therapy.
10. Must be willing to report baseline and required patient-reported outcomes and use the Dieta app for monitoring stool changes.
11. For a female subject of childbearing potential, must have documentation of a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 1. All women are considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 2 years) or documented to be surgically sterile (bilateral tubal ligation or hysterectomy).
12. Sexually active subjects must use a highly effective method of contraception during the study and for at least 90 days after completion of study drug dosing.

    1. A highly effective method of birth control is defined as one that results in a low failure rate (i.e., < 1% per year) when used consistently and correctly, such as condom + diaphragm, condom + spermicide, diaphragm + spermicide, or intrauterine device (IUD) with documented failure rate of < 1% per year, or oral/injectable/implanted hormonal contraceptives used in combination with an additional barrier method.
    2. Males should refrain from donating sperm during the study and for 90 days after completion of study drug.

Exclusion Criteria:

1. Any previous gastrointestinal surgery, except uncomplicated appendectomy or cholecystectomy.
2. Any of the included cancer cohorts where active malignancy causes direct extension/invasion of the GI tract from local spread or distant metastasis.
3. Current, active, untreated brain metastases.
4. History of fecal incontinence/impaction; irritable bowel syndrome; inflammatory bowel disease; intestinal obstruction; GI or pelvic disorders known to affect bowel transit, produce GI obstruction, or contribute to bowel dysfunction; fecal impaction requiring medical intervention within 1 month of enrollment.
5. Subject is unable to eat, drink, take, or hold down oral medications.
6. Use of buprenorphine, alvimopan, naltrexone, methylnaltrexone, naloxone, lubiprostone, linaclotide, or tapentadol therapy within 14 days before enrollment and inability or unwillingness to discontinue use until the end of the study.
7. Receipt of strong inhibitors of CYP3A4 (e.g., antifungal azoles, grapefruit juice) or strong inducers of CYP3A4 (e.g., rifampin or carbamazepine), including any herbal medications such as St. John's Wort, within the last 14 days or 5 half-lives, whichever is longer, prior to study drug administration.
8. Receipt of inhibitors of p-glycoprotein (P-gp) within the last 14 days prior to study drug administration.
9. Receipt of anti-VEGF therapies (i.e. bevacizumab) within the last 30 days prior to study drug administration.
10. Subjects with clinically significant abnormal ECG at screening or before randomization in the opinion of the Investigator, or a QTc > 470 msec (per Fridericia's correction).
11. Presence of unstable diseases, in the opinion of the Investigator, such as cardiovascular (e.g., acute myocardial infarction or acute coronary syndrome < 3 month history), respiratory (e.g., requires oxygen), gastrointestinal (e.g., symptomatic diverticulitis, irritable bowel syndrome [IBS], etc.), endocrine (e.g., uncontrolled diabetes or A1c > 10%), hematologic, neurologic, psychiatric (e.g., schizophrenia, unstable anxiety disorder, acute psychosis, depression with suicidal ideation, etc.), or any other significant conditions that may affect subject assessment.
12. Any other condition which, in the opinion of the investigator, could confound or interfere with evaluation of safety, efficacy, or tolerability of the investigational drug, or prevent compliance with the study protocol.
13. Women who are pregnant, breastfeeding, or of childbearing potential without the use of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (including complete response and partial response) | 43 days
  Calculate objective response rate (including complete response and partial response) at day 43 based on RECIST 1.1 (and PCWG3 for prostate cohort) criteria.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 43 days
  Determine the disease control rate (DCR) (defined as the percentage of patients who achieve a CR, partial response, or stable disease) and progression-free survival based on RECIST 1.1 (and PCWG3 for prostate cohort) criteria.
Impact on ctDNA | 43 days
  Assess the change in cancer-specific tumor markers (if applicable) and ctDNA from baseline to day 43.
Impact on bowel function | 43 days
  Evaluate the bowel function and patient-reported outcomes related to constipation associated with use of axelopran.
Impact on systemic inflammation | Day 43
  Conduct correlative studies on systemic inflammation as assessed through routine collection of albumin, neutrophil/lymphocyte ratios, and inflammatory markers (ESR, CRP, IL-6, and TNFa).

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Zylla, MD, MS, Principal Investigator — HealthPartners Institute Cancer Research Center
Locations (2):
- United States (2):
  - HealthPartners Frauenshuh Cancer Research Center, Saint Louis Park, Minnesota
  - HealthPartners Cancer Center at Regions Hospital, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Yes